CLINICAL TRIAL: NCT06785675
Title: Assessing Short-term Treatment Satisfaction and Quality of Life in Patients With Hidradenitis Suppurativa Initiated on Secukinumab in Routine Clinical Practice in the United Arab Emirates: ILLUMINATE-HS, a Prospective Patient Surve
Brief Title: Assessing Short-term Treatment Satisfaction and Quality of Life in Patients With Hidradenitis Suppurativa Initiated on Secukinumab.
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457AAE02
Record Dates: First submitted 2024-11-27; First posted 2025-01-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Secukinumab: Patients who are newly initiated on treatment with Secukinumab
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — This is an observational study. There is no treatment allocation.

SUMMARY:
This study will be conducted to address the lack of concrete data on the impact of pharmaceutical intervention on short-term patient satisfaction and quality of life (QoL) in patients with Hidradenitis Suppurativa (HS) in real-world settings, especially in the Gulf Region.

DETAILED DESCRIPTION:
This is a 24-week longitudinal single-arm prospective study based on data collected from EMRs along with patient-reported outcomes questionnaires (TSQM and DLQI) to evaluate patient-reported satisfaction and early quality of life experiences among HS patients who are newly initiated on Secukinumab. We will be using questionnaires at baseline and at week 24 to report on pre-defined outcomes in a representative HS population across the United Arab Emirates. The data will be collected using an electronic Case Report Form (eCRF) from both data sources (Electronic Medical Report and Questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a confirmed diagnosis of active moderate to severe HS (Hurley Score 2-3)
* Male or Female adult patients ≥ 18 years of age at the time of data collection
* Patient newly initiated on Secukinumab (first dose to coincide within 1 month of the signature of the informed consent)
* Patients with a diagnosis of HS who are currently using antibiotics/ have undergone surgery or not as part of their routine clinical management are eligible for inclusion.
* Patients with a diagnosis of HS who have a history of previous treatment with Adalimumab or any other anti-TNF agent as part of their routine clinical management or biologic naïve are eligible for inclusion.
* Agreed to sign an informed consent to be able to fill in the questionnaires.

Exclusion Criteria:

* Patients not fulfilling any of the abovementioned inclusion criteria.
* Patient's refusal to be included in the study or refusal to sign the informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hidradenitis Suppurativa who are newly initiated on Secukinumab, across the United Arab Emirates.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The absolute scores of each of the 4 domains of the Treatment Satisfaction Questionnaire for Medication (TSQM) questionnaire | At Week 24
  TSQM scoring is calculated by domain, and each domain score is computed by summing the individual TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100, with higher scores indicating higher patient satisfaction.
  4 Domains:
  Effectiveness Side Effects Convenience Global Satisfaction

SECONDARY OUTCOMES:
Change from baseline of the Dermatology Life Quality Index (DLQI) Questionnaire | Baseline, Week 24
  DLQI is a questionnaire designed to measure the impact of skin conditions on a patient's health-related quality of life. It contains 10 simple, self-administered questions. Focuses on the past week's experiences related to the skin condition. Each question uses a 4-point Likert scale: "Not at all," "A little," "A lot," "Very much."
Change from baseline in the Numerical Rating Scale (NRS) | Baseline, Week 24
  The NRS is commonly used for measuring pain intensity and is well validated. It is scored from 0-10 (0 meaning no pain and 10 meaning the worst pain imaginable).
Age (years) | Baseline
  Characteristics of Hidradenitis Suppurativa (HS) patients started on Secukinumab
Gender (male/female) | Baseline
  Characteristics of HS patients started on Secukinumab
Ethnicity | Baseline
  Characteristics of HS patients started on Secukinumab
Weight (kilogram) | Baseline
  Characteristics of HS patients started on Secukinumab
Height (meters) | Baseline
  Characteristics of HS patients started on Secukinumab
Socio-economic status | Baseline
  Characteristics of HS patients started on Secukinumab
Smoking status | Baseline
  Characteristics of HS patients started on Secukinumab
Duration of the disease (time since diagnosis) | Baseline
  Characteristics of HS patients started on Secukinumab
Previous HS-related treatment | Baseline
  Characteristics of HS patients started on Secukinumab
Time since diagnosis to start of the first treatment, and from time since diagnosis to start of Secukinumab | Baseline
  Characteristics of HS patients started on Secukinumab
Hurley Stage | Baseline
  Characteristics of HS patients started on Secukinumab
Number of inflammatory nodules, number of abscesses, and fistulas | Baseline
  Characteristics of HS patients started on Secukinumab
Previous HS-related surgeries | Baseline
  Characteristics of HS patients started on Secukinumab
Previous use of biologic treatment | Baseline
  Characteristics of HS patients started on Secukinumab
Previous and current use of antibiotics treatment | Baseline
  Characteristics of HS patients started on Secukinumab

CONTACTS AND LOCATIONS:
Locations (4):
- United Arab Emirates (4):
  - Novartis Investigative Site, Al Ain Abu Dhabi, United Arab Emirates
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Ras al-Khaimah
  - Novartis Investigative Site, Sharjah city